CLINICAL TRIAL: NCT03004183
Title: Phase II Window of Opportunity Trial of Stereotactic Body Radiation Therapy and In Situ Oncolytic Virus Therapy in Metastatic Triple Negative Breast Cancer and Metastatic Non-Small Cell Lung Cancer Followed by Pembrolizumab
Brief Title: SBRT and Oncolytic Virus Therapy Before Pembrolizumab for Metastatic TNBC and NSCLC
Acronym: STOMP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Jenny C. Chang, MD, Director of the Houston Methodist Cancer Center, The Methodist Hospital Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00015649
Record Dates: First submitted 2016-12-20; First posted 2016-12-28 (Estimated); Results first posted 2023-01-25 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-08

CONDITIONS: Metastatic Non-small Cell Lung Cancer; Metastatic Triple-negative Breast Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms | interventions — Valacyclovir; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): ADV/HSV-tk (5 x 1011 virus particles) in a 2-mL total volume will be injected intratumorally on Day 0.
  Valacyclovir will be orally administered at a dose of 2 g three times daily for 14 days from Day 1 to Day 15.
  SBRT of 30 Gy (6 Gy X 5 fractions) will be administered over 2 weeks from Day 2 to Day 16.
  Pembrolizumab (200 mg) will be administered intravenously over 30 minutes every 3 weeks starting on Day 17 and continuing until disease progression, unacceptable toxicity, or up to 24 months in patients without disease progression.
  Interventions: Biological: ADV/HSV-tk; Drug: Valacyclovir; Radiation: SBRT; Drug: Pembrolizumab

INTERVENTIONS:
Biological: ADV/HSV-tk — Replication-defective recombinant adenovirus vector
Drug: Valacyclovir — Prodrug of the antiviral drug acyclovir
  Other Names: valacyclovir hydrochloride
Radiation: SBRT — Low-dose SBRT
Drug: Pembrolizumab — Humanized immunoglobulin G4 anti-programmed death-1 (PD-1) monoclonal antibody
  Other Names: Keytruda

SUMMARY:
This is a Phase II trial to determine the efficacy and safety of stereotactic body radiation therapy (SBRT) and in situ oncolytic virus therapy used as a window of opportunity treatment before pembrolizumab in patients with metastatic triple negative breast cancer (TNBC) and metastatic non-small cell lung cancer (NSCLC). In situ oncolytic virus therapy will consist of adenovirus-mediated expression of herpes simplex virus thymidine kinase (ADV/HSV-tk) plus valacyclovir therapy.

DETAILED DESCRIPTION:
This is a Phase II trial to determine the efficacy and safety of stereotactic body radiation therapy (SBRT) and in situ oncolytic virus therapy used as a window of opportunity treatment before pembrolizumab in patients with metastatic triple negative breast cancer (TNBC) and metastatic non-small cell lung cancer (NSCLC). In situ oncolytic virus therapy will consist of adenovirus-mediated expression of herpes simplex virus thymidine kinase (ADV/HSV-tk) plus valacyclovir. Male and female patients aged ≥ 18 years with histologically confirmed locally advanced or metastatic TNBC that has relapsed on or is refractory to 1 or more lines of standard of care therapy or histologically or cytologically confirmed metastatic NSCLC that is immunotherapy and chemotherapy naïve or previously treated with 1 cycle of platinum-containing chemotherapy are eligible to participate in the study. ADV/HSV-tk (5 x 1011 viral particles) in a 2-mL total volume will be injected intratumorally on Day 0 of the study. Valacyclovir will be orally administered at a dose of 2 g three times daily for 14 days. Valacyclovir treatment will be administered 24 hours after the gene vector injection from Day 1 to Day 15 of the study. SBRT of 30 gray (Gy; 6 Gy X 5 fractions) will be administered over 2 weeks from Day 2 to Day 16 of the study. Pembrolizumab (200 mg) will be administered intravenously over 30 minutes every 3 weeks starting on Day 17 of the study and continuing until disease progression, unacceptable toxicity, or up to 24 months in patients without disease progression. The primary endpoint will be the objective response rate of ADV/HSV-tk + valacyclovir therapy in combination with SBRT used as a window of opportunity treatment before pembrolizumab in patients with metastatic TNBC and metastatic NSCLC. RECIST 1.1 will be used to assess treatment response. Secondary endpoints will include a) clinical benefit rate; b) duration of response; c) overall survival and progression-free survival rates; d) toxicity (toxicity will be defined as any treatment-related death or any ≥ grade 3 toxicity excluding alopecia and constitutional symptoms as assessed by the NCI CTCAE v4.03); and e) antitumor activity of ADV/HSV-tk plus valacyclovir therapy in combination with SBRT used as a window of opportunity treatment before pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent/assent for the trial.
2. Male or female aged ≥18 years on the day of informed consent signing.
3. Histologically confirmed locally advanced or metastatic TNBC that has relapsed on or is refractory to standard of care therapy OR histologically or cytologically confirmed metastatic NSCLC that is immunotherapy and chemotherapy naïve or previously treated with 1 cycle of platinum-containing chemotherapy. Epidermal growth factor receptor (EGFR)/anaplastic lymphoma kinase (ALK) mutation-negative NSCLC patients and NSCLC patients with EGFR or ALK genomic tumor aberrations that have failed FDA-approved targeted therapy for these aberrations will be eligible for enrollment in the study.
4. Measurable disease based on RECIST 1.1, a target lesion of suitable diameter (at least 1 cm) for SBRT, and a non-target lesion (visceral metastatic lesion) at least 1 cm in diameter for abscopal effect evaluation.
5. Willing to provide biopsy tissues as required by the study.
6. Eastern Cooperative Oncology Group performance status of 0 or 1.
7. Adequate organ function as defined by the following laboratory values:

   * Absolute neutrophil count ≥1,500/µL (without granulocyte colony stimulating factor support within 14 days of assessment)
   * Platelets ≥100,000/µL
   * Hemoglobin ≥8 g/dL or ≥5.6 mmol/L without transfusion or erythropoietin dependency (within 7 days of assessment)
   * White blood cell count >2,500/µL and <15,000/µL
   * Lymphocyte count ≥500/µL
   * Serum creatinine <2 X upper limit of normal (ULN)
   * Serum total bilirubin ≤1.0 X ULN (Subjects with known Gilbert's disease who have serum bilirubin level ≤3 X ULN may be enrolled)
   * Asparate transaminase and alanine transaminase ≤2.5 X ULN with normal alkaline phosphatase (≤5 X ULN for subjects with liver metastases) OR ≤1.5 X ULN in conjunction with alkaline phosphatase >2.5 X ULN
   * Albumin >2.5 mg/dL
   * International normalized ratio or prothrombin time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or activated partial thromboplastin time (aPTT) is within therapeutic range of intended use of anticoagulants
   * aPTT ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
8. Life expectancy ≥ 6 months.
9. ≥ 4 weeks since any major surgery, completion of radiation therapy, or completion of all prior systemic anticancer therapy (adequately recovered from the acute toxicities of any prior therapy).
10. Female subjects of childbearing potential should have a negative serum pregnancy (beta-human chorionic gonadotropin) within 7 days prior to receiving the first dose of the trial treatment and should not be lactating.
11. Female subjects of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study therapy.
12. Male subjects of childbearing potential must agree to use an adequate method of contraception for the course of the study through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Unwilling or unable to comply with the study protocol.
2. Subjects for who bone metastases are the only available non-target lesions for abscopal effect evaluation.
3. Subjects with tumors for which SBRT is not considered appropriate standard therapy. This includes subjects with target lesions less than 1 cm in diameter and those with large central lung lesions.
4. Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of trial treatment.
5. Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
6. Known history of active tuberculosis (Bacillus Tuberculosis).
7. Known or suspected hypersensitivity to pembrolizumab or any of its excipients or any component of the proposed regimen (gene vector/valacyclovir).
8. Known gallbladder or bile duct disease (i.e., infection or cholecystitis) or acute or chronic pancreatitis.
9. Eastern Cooperative Oncology Group performance status of ≥2 or oxygen dependence (e.g., advanced chronic obstructive pulmonary disease).
10. Inability to swallow food or any condition of the upper gastrointestinal tract that precludes administration of oral medications (valacyclovir).
11. Congestive heart failure: New York Association class III or IV heart failure or unstable angina.
12. Sustained or clinically significant cardiac arrhythmias including sustained ventricular tachycardia, ventricular fibrillation, clinically significant bradycardia, advanced heart block (Mobitz II or higher atrioventricular nodal block), prolonged corrected QT interval (longer than 470 milliseconds), or history of acute myocardial infarction.
13. Concomitant disease(s) that could prolong QT such as autonomic neuropathy (caused by diabetes or Parkinson's disease), human immunodeficiency virus (HIV), cirrhosis, uncontrolled hypothyroidism, or cardiac failure.
14. History of syncope or family history of idiopathic sudden death.
15. Targeted small molecule therapy or monoclonal antibody or radiation therapy within 3 weeks prior to study Day 0 or has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

    - Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
16. Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
17. Known active central nervous system metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 4 weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability.
18. Active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
19. History of (non-infectious) pneumonitis that required steroids or current pneumonitis.
20. Active infection requiring systemic therapy.
21. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
22. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
23. Pregnant or breastfeeding, expecting to conceive or father children within the projected duration of the trial, starting with the prescreening or screening visit through 120 days after the last dose of trial treatment, or is unwilling to practice an effective method of birth control. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to administration of trial treatment.
24. Prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent (TNBC cohort only).
25. Prior treatment with immunomodulatory therapy or immunotherapy (TNBC cohort only).
26. Prior treatment with gene vector therapy.
27. Received prior systemic cytotoxic chemotherapy for metastatic disease (NSCLC cohort).
28. Known history of HIV (HIV 1/2 antibodies).
29. History of liver disease such as cirrhosis or known active hepatitis B (e.g., hepatitis B surface antigen reactive) or hepatitis C (e.g., hepatitis C virus RNA [qualitative] is detected).
30. History of or current alcohol misuse/abuse within the past 12 months.
31. Major surgery within 4 weeks prior to study enrollment.
32. Received a live vaccine within 30 days of planned start of trial therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2024-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Chang, MD, Principal Investigator — Houston Methodist Cancer Center
Locations (1):
- Houston Methodist Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data and materials on human subjects will be shared with other eligible investigators through appropriate means in accordance with the NIH policy on Sharing Research Data (NIH Guide, February 26, 2003). Data will be also shared with the funding agency and regulatory agencies as required. Data will be shared with other investigators within the limits of HIPAA and other patient confidentiality requirements. This will generally require removal of all patient identifiers for all source documents and the use of arbitrarily assigned one-way identifiers. In some cases, requestors will be asked to sign a formal data sharing agreement that will provide for a commitment to use data only for research purposes and not to identify individuals, keep the data secure, and destroy or return data after analyses are complete. Prior approval will be obtained from collaborating investigators, research sponsors, and/or other stake-holders before sharing if proprietary information or products are involved.
Supporting Information: Study Protocol
Time Frame: During and/or after result submission.
Access Criteria: The study protocol will be included on clinicaltrials.gov

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 57 overall participants (28 TNBC and 29 NSCLS)
Pre-assignment Details: The Triple Negative Breast Cancer (TNBC) patients with histologically confirmed locally advanced or metastatic TNBC that has relapsed or is refractory to ≥1 lines of standard of care therapy. The Non-Small Cell Lung Cancer (NSCLC) cohort will include male & female patients with confirmed metastatic NSCLC that is immunotherapy naïve or previously treated with a maximum of 1 immunotherapy regimen & chemotherapy naïve or previously treated with 1 cycle of platinum-containing chemotherapy.
Groups:
- Single Arm: ADV/HSV-tk (5 x 1011 virus particles) in a 2-mL total volume will be injected intratumorally on Day 0.
  Valacyclovir will be orally administered at a dose of 2 g three times daily for 14 days from Day 1 to Day 15.
  SBRT of 30 Gy (6 Gy X 5 fractions) will be administered over 2 weeks from Day 2 to Day 16.
  Pembrolizumab (200 mg) will be administered intravenously over 30 minutes every 3 weeks starting on Day 17 and continuing until disease progression, unacceptable toxicity, or up to 24 months in patients without disease progression.
  ADV/HSV-tk: Replication-defective recombinant adenovirus vector
  Valacyclovir: Prodrug of the antiviral drug acyclovir
  SBRT: Low-dose SBRT
  Pembrolizumab: Humanized immunoglobulin G4 anti-programmed death-1 (PD-1) monoclonal antibody
Period: Overall Study
Arm/Group | Single Arm
Started | 57
TNBC | 28
NSCLC | 29
Completed | 7 (1 TNBC and 6 NSCLC)
Not Completed | 50
Not completed — Adverse Event | 7
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 40
Not completed — Withdrawal by Subject | 1
Not completed — COVID-19 | 1

BASELINE CHARACTERISTICS:
Population: There are 57 total patients enrolled in this trial, the results are based on a total of 56 patients (28 TNBC and 28 NSCLC evaluable patients).
Arm/Group | Single Arm
Number analyzed (Participants) | 56
Age, Categorical [Count of Participants; unit: Participants] — Population: The results are distributed based on a total of 56 patients, 28 TNBC and 28 NSCLC evaluable patients.
  Participants
    Overall: <=18 years | 0
    Overall: Between 18 and 65 years | 32
    Overall: >=65 years | 24
    TNBC: number analyzed (Participants) | 28
    TNBC: <=18 years | 0
    TNBC: Between 18 and 65 years | 24
    TNBC: >=65 years | 4
    NSCLC: number analyzed (Participants) | 28
    NSCLC: <=18 years | 0
    NSCLC: Between 18 and 65 years | 8
    NSCLC: >=65 years | 20
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The results are distributed based on a total of 56 patients, 28 TNBC and 28 NSCLC evaluable patients.
  Participants
    Overall: Female | 40
    Overall: Male | 16
    TNBC: number analyzed (Participants) | 28
    TNBC: Female | 28
    TNBC: Male | 0
    NSCLC: number analyzed (Participants) | 28
    NSCLC: Female | 12
    NSCLC: Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The results are distributed based on a total of 56 patients, 28 TNBC and 28 NSCLC evaluable patients.
  Participants
    Overall: Hispanic or Latino | 4
    Overall: Not Hispanic or Latino | 52
    Overall: Unknown or Not Reported | 0
    TNBC: number analyzed (Participants) | 28
    TNBC: Hispanic or Latino | 3
    TNBC: Not Hispanic or Latino | 25
    TNBC: Unknown or Not Reported | 0
    NSCLC: number analyzed (Participants) | 28
    NSCLC: Hispanic or Latino | 1
    NSCLC: Not Hispanic or Latino | 27
    NSCLC: Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The results are distributed based on a total of 56 patients, 28 TNBC and 28 NSCLC evaluable patients.
  Participants
    Overall: American Indian or Alaska Native | 0
    Overall: Asian | 6
    Overall: Native Hawaiian or Other Pacific Islander | 0
    Overall: Black or African American | 9
    Overall: White | 41
    Overall: More than one race | 0
    Overall: Unknown or Not Reported | 0
    TNBC: number analyzed (Participants) | 28
    TNBC: American Indian or Alaska Native | 0
    TNBC: Asian | 5
    TNBC: Native Hawaiian or Other Pacific Islander | 0
    TNBC: Black or African American | 5
    TNBC: White | 18
    TNBC: More than one race | 0
    TNBC: Unknown or Not Reported | 0
    NSCLC: number analyzed (Participants) | 28
    NSCLC: American Indian or Alaska Native | 0
    NSCLC: Asian | 1
    NSCLC: Native Hawaiian or Other Pacific Islander | 0
    NSCLC: Black or African American | 4
    NSCLC: White | 23
    NSCLC: More than one race | 0
    NSCLC: Unknown or Not Reported | 0
TNBC and NSCLC patient distribution [Count of Participants; unit: Participants]
  TNBC | 28
  NSLC | 28

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: The objective response rate (ORR) of ADV/HSV-tk plus (+) valacyclovir therapy in combination with SBRT used as a window of opportunity treatment before pembrolizumab in patients with metastatic TNBC and metastatic NSCLC. Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 will be used to assess treatment response. Modified immune-related response criteria (irRC; derived from RECIST 1.1) will also be documented.
Time Frame: 30 days after the last dose of pembrolizumab until disease progression, initiating a non-study cancer treatment, withdrawing consent, or becoming lost to follow-up. Median duration of follow-up was 8.3 months (95% CI 3.0-10.1 months).
Population: A total of 56 patient's data was analyzed, 28 patients with mTNBC and 28 patients with NSCLC.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 56
Participants
  Overall: Complete Response | 4
  Overall: Partial Response | 7
  Overall: Stable Diseases | 13
  Overall: Progressive Disease | 32
  TNBC: number analyzed (Participants) | 28
  TNBC: Complete Response | 2
  TNBC: Partial Response | 1
  TNBC: Stable Diseases | 3
  TNBC: Progressive Disease | 22
  NSCLC: number analyzed (Participants) | 28
  NSCLC: Complete Response | 2
  NSCLC: Partial Response | 6
  NSCLC: Stable Diseases | 10
  NSCLC: Progressive Disease | 10

2. Secondary Outcome: Duration of Response
Description: Duration of response to ADV/HSV-tk plus valacyclovir therapy in combination with SBRT followed by pembrolizumab
Time Frame: as for outcome 1
Population: Median duration of response from last line of treatment (range), months
Measure: Median (Full Range); unit: Months
Arm/Group | Single Arm
Number analyzed (Participants) | 56
Months
  TNBC: number analyzed (Participants) | 28
  TNBC | 2 [1 to 7]
  NSCLC: number analyzed (Participants) | 28
  NSCLC | 5.5 [0 to 13]

3. Secondary Outcome: Overall Survival Rate
Description: Overall survival (OS) rate in subjects receiving ADV/HSV-tk plus valacyclovir therapy in combination with SBRT followed by pembrolizumab. OS is the time (measured in months) from intratumoral viral injection to death or last date of contact.
Time Frame: After confirmed disease progression or starts a new therapy, the subject moves into the Survival Follow-up to be contacted every 12 weeks to assess for survival status until death, withdrawal, or end of study. Median duration of follow-up was 8.3 months.
Population: Median overall survival for all patient and for patients with clinical benefit
Measure: Median (Full Range); unit: Months
Arm/Group | Single Arm
Number analyzed (Participants) | 56
Months
  TNBC: number analyzed (Participants) | 28
  TNBC | 6.6 [0 to 50]
  NSCLC: number analyzed (Participants) | 28
  NSCLC | 12.9 [0 to 32]

4. Secondary Outcome: Number of Participants With Treatment-related Adverse Events
Description: To document the toxicities associated with ADV/HSV-tk + valacyclovir therapy in combination with SBRT used as a window of opportunity treatment before pembrolizumab in patients with metastatic TNBC and metastatic NSCLC. Toxicity will be defined as the number of participants with any treatment-related death or any ≥ Grade 3 hematological toxicity excluding alopecia and constitutional symptoms, as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.03.
Time Frame: Adverse Events (AEs) and Serious Adverse Events (SAEs) will be captured from the time of informed consent signing up to 30 days after the final dose of pembrolizumab, (up to 24 months of treatment for patients without disease progression).
Population: The results are distributed based on a total of 56 patients, 28 TNBC and 28 NSCLC evaluable patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 56
Participants
  Total with Related SAE | 2
  TNBC: number analyzed (Participants) | 28
  TNBC | 2
  NSCLC: number analyzed (Participants) | 28
  NSCLC | 0

5. Secondary Outcome: Antitumor Activity
Description: Measure the antitumor activity as assessed by RECIST 1.1. Modified immune-related response criteria will also be documented.
Time Frame: 30 days after the last dose of pembrolizumab
Population: At this point in the data analysis has not been completed, information will be updated as it becomes available.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 56
Participants
  Overall: Complete Response | 4
  Overall: Partial Response | 7
  Overall: Stable Diseases | 13
  Overall: Progressive Disease | 32
  TNBC: number analyzed (Participants) | 28
  TNBC: Complete Response | 2
  TNBC: Partial Response | 1
  TNBC: Stable Diseases | 3
  TNBC: Progressive Disease | 22
  NSCLS: number analyzed (Participants) | 28
  NSCLS: Complete Response | 2
  NSCLS: Partial Response | 6
  NSCLS: Stable Diseases | 10
  NSCLS: Progressive Disease | 10

6. Secondary Outcome: Clinical Benefit Rate
Description: Clinical benefit rate of ADV/HSV-tk plus valacyclovir therapy in combination with SBRT followed by pembrolizumab
Time Frame: as for outcome 1
Population: The Clinical Benefit Rate measured as Complete Response plus Partial Response plus Stable Disease
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 56
Participants
  Overall | 24
  TNBC: number analyzed (Participants) | 28
  TNBC | 6
  NSCLC: number analyzed (Participants) | 28
  NSCLC | 18

7. Secondary Outcome: Progression-free Survival in Months
Description: To determine the progression-free survival (PFS) of ADV/HSV-tk + valacyclovir therapy in combination with SBRT used as a window of opportunity treatment before pembrolizumab in patients with metastatic TNBC and metastatic NSCLC as measured in months and defined the number of months a patient remains free from disease progression.
Time Frame: 30 days after the last dose of pembrolizumab until disease progression, initiating a non-study cancer treatment, withdrawing consent, or becoming lost to follow-up.
Population: Median duration of progression free response from last line of treatment (range), months
Measure: Median (Full Range); unit: months
Arm/Group | Single Arm
Number analyzed (Participants) | 56
months
  TNBC: number analyzed (Participants) | 28
  TNBC | 2.5298 [1.05 to 48.53]
  NSCLC: number analyzed (Participants) | 28
  NSCLC | 7.4 [5.1 to 9.6]

8. Other Pre Specified Outcome: Computed Tomography-based Response of a Non-target Lesion
Description: Measure the computed tomography-based response (RECIST 1.1) of a non-target lesion to ADV/HSV-tk plus valacyclovir therapy in combination with SBRT followed by pembrolizumab
Time Frame: baseline and 30 days after the last dose of pembrolizumab
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in Immunohistochemical Expression of Tumor-infiltrating Lymphocytes in Tumor Biopsy Tissues
Description: Measure the change in immunohistochemical expression of tumor-infiltrating lymphocytes in tumor biopsy tissues in response to ADV/HSV-tk plus valacyclovir therapy in combination with SBRT followed by pembrolizumab
Time Frame: baseline and 30 days after the last dose of pembrolizumab
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: AEs and SAEs will be captured from the time of informed consent signing up to 30 days after the final dose of pembrolizumab. Study treatment-related SAEs and any study patient death occurring beyond 30 days after the last dose of pembrolizumab should also be reported. Patients will be treated until disease progression, unacceptable toxicity, or up to 24 months in subjects without disease progression.
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 17/56
Serious Adverse Events (participants affected / at risk) | 29/56
Other Adverse Events (participants affected / at risk) | 28/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=56)
Intractable pain, back pain, hip pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2)
Atrial fibrillation with rapid ventricular response (Cardiac disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (4)
colitis (Gastrointestinal disorders) | 1 (1)
Malnutrition, Hypercalcemia and Weakness (Metabolism and nutrition disorders) | 3 (4)
Kidney Injury and/or Infection (Renal and urinary disorders) | 4 (6)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Skin rash (Skin and subcutaneous tissue disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=56)
Anemia (Blood and lymphatic system disorders) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 7 (7)
Fatigue (General disorders) | 12 (12)
Activated partial thromboplastin time prolonged (Investigations) | 3 (10)
Weight Loss (Investigations) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-25): https://cdn.clinicaltrials.gov/large-docs/83/NCT03004183/Prot_SAP_000.pdf